CLINICAL TRIAL: NCT00734357
Title: Comparative Investigation of Intravenously Administered Omnipaque and Isovue: Effects on Serum Creatinine Concentration in Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Mahmoud Al-Hawary, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00019769
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Kidney Disease
Keywords: contrast; ct; cat scan; kidney; nephrotoxicity; Computerized Emission Tomography
MeSH Terms: conditions — Kidney Diseases

ARMS (2):
- Isovue Arm (Experimental): Subjects with a clinically scheduled CT examination will be given the contrast Isovue. The investigators of this study will determine which contrast medication subjects will receive using randomization.
  Interventions: Procedure: Blood work
- Omnipaque Arm (Experimental): Subjects with a clinically scheduled CT examination will be given the contrast Omnipaque. The investigators of this study will determine which contrast medication subjects will receive using randomization
  Interventions: Procedure: Blood work

INTERVENTIONS:
Procedure: Blood work — Prior to having the clinically scheduled CT examination the subject will have blood work drawn. This blood work will give the investigators a baseline value of the basic kidney function of the subject. They will then have blood work done again at 2 days and again at 3 days following the CT examination. Some patients, based on their blood work obtained at 2 and 3 days after the CT examination, will be asked to have blood work performed at 7 days after their CT examination.

SUMMARY:
The purpose of this study is to determine if one CT contrast agent (medication injected into a vein; used in CT examinations to help produce clearer images) is safer to use than another. This study will compare the safety of two widely-used, U.S. FDA approved contrast agents, Isovue and Omnipaque. The investigators hypothesize that there is no significant difference in the rates of contrast-induced nephrotoxicity (CIN) between these agents when the overall population consists of low-risk patients.

DETAILED DESCRIPTION:
For patients without known kidney disease, it is exceptionally rare for the administration of CT contrast agents to injure the kidneys, and those rare injuries that do occur are almost always temporary (a week or two) and heal. Indeed, significant injuries are so rare that the kidney function in patients is not routinely checked after they receive CT contrast agents. There are many brands of contrast media in common use across the United States, and it has been thought in the past that all are similarly low in risk. The purpose of this study is to examine whether two different contrast materials might differ in their risk to the kidneys. We will perform a direct comparison of Omnipaque-300 (iohexol, 300 mg I/ml) and Isovue-300 (Iopamidol, 300 mg I/ml) low osmolality contrast agents to determine their relative CIN rates (as measured by serum creatinine concentration) in low-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Patients referred for a contrast-enhanced CT examination. Such contrast- enhanced CT examinations include, but are not limited to, certain examinations of the head, neck, chest, abdomen, pelvis, etc.

Exclusion Criteria:

* Patients less than age of 18 years of age
* Pregnant patients
* Patients unable to provide written informed consent
* Patients in whom there are contraindications to the administration of intravenous contrast material (as detailed in out Department of Radiology intravenous contrast material use guidelines), including renal contraindications (such as a University of Michigan laboratory record of most recent serum creatinine concentration of >1.5 mg/dl or an estimated glomerular filtration rate (EGFR) <60 ml/min); if no serum creatinine is available, patients will be receive contrast material based on departmental guidelines
* Patients who are undergoing therapy with agents purported to reduce the risk of CIN (such as acetylcysteine, theophylline, or intravenous hydration)
* Patients who are unable to provide the follow-up serum creatinine concentration measurements
* Patients undergoing CT examinations that utilize a higher concentration of iodine (for example, 370 mg I/ml contrast material)
* Patients who have experienced allergic-like reactions to contrast; including patients who receive corticosteroid/antihistamine premedication to reduce the risk of an acute allergic-like reaction
* Patients who do not receive the study criterion for dose of contrast material; and patients in whom a contrast extravasation of more than 5 ml occurs (so that it is not possible to determine how much contrast material the patient received as a direct intravenous injection)
* Patients participating in other investigational drug, contrast material, or device trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the change in serum creatinine concentration from the baseline obtained immediately prior to contrast administration. | 48 and 72 hours from the baseline exam

SECONDARY OUTCOMES:
We will also identify the number of patients in each group who develop CIN. Two separate CIN definitions will be utilized, including a rise in serum creatinine of 0.5 mg/dl from baseline and a rise in serum creatinine of 25% or greater from baseline. | 48 and 72 hours from the baseline exam

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States